CLINICAL TRIAL: NCT01465230
Title: Maintenance Therapy With Lenalidomide Following Bendamustine and Rituximab Induction Therapy for Chronic Lymphocytic Leukemia
Brief Title: Maintenance Therapy: Lenalidomide Following Bendamustine and Rituximab Induction Therapy for Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was unsuccessful in enrolling the target number of subjects during the funding period.
Sponsor: Yale University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1105008515
Record Dates: First submitted 2011-10-28; First posted 2011-11-04 (Estimated); Results first posted 2014-10-23 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; maintenance therapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lenalidomide (Experimental): Maintenance treatment with lenalidomide following induction treatment with bendamustine and rituximab.
  Interventions: Drug: Maintenance lenalidomide

INTERVENTIONS:
Drug: Maintenance lenalidomide — Daily maintenance treatment, oral lenalidomide

SUMMARY:
This study will determine whether or not Lenalidomide improves effectiveness of treatment for chronic lymphocytic leukemia following chemotherapy with two drugs commonly used to treat the disease (bendamustine and rituximab).

ELIGIBILITY:
Inclusion Criteria:

* Previous induction treatment with bendamustine and rituximab
* 18 or more years of age
* chronic lymphocytic leukemia
* ECOG performance status less than or equal to 2
* Absolute neutrophile count more than 1,000
* Platelet count more than 70,000

Exclusion Criteria:

* Serious medical condition that would prevent treatment with lenalidomide
* Evidence of tumor lysis syndrome
* Any prior treatment with lenalidomide

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terri L Parker, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 36 months
Population: Participants withdrew from study before primary outcome could be measured
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the length of the study (approximately 1 year and 1/2)
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=2)
Deep Vein Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1
Decreased Platlets (Blood and lymphatic system disorders) | 1
Sciatica Pain (Musculoskeletal and connective tissue disorders) | 1
Bilateral Hand Spasticity (Musculoskeletal and connective tissue disorders) | 1
Decreased ANC (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Decreased Calcium (Blood and lymphatic system disorders) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Decreased Neutrophil Count (Blood and lymphatic system disorders) | 1
Syncope (General disorders) | 1
Right Groin Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes